CLINICAL TRIAL: NCT05596786
Title: Evaluation de l'efficacité et de la sécurité du Rituximab Chez Les Patients Avec Une Pneumopathie Interstitielle Diffuse Progressive Avec Composante Inflammatoire : Essai Clinique randomisé Multicentrique en Double Insu Contre Placebo
Brief Title: Evaluation of Efficacy and Safety of Rituximab in Patients With Progressive Interstitial Lung Disease (ILD) With Inflammatory Component: a Multicentre Double-blind Placebo-controlled Randomized Trial
Acronym: EvER-ILD2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DR210299
Record Dates: First submitted 2022-10-19; First posted 2022-10-27 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Lung Diseases
MeSH Terms: conditions — Lung Diseases | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rituximab (Experimental)
  Interventions: Drug: Rituximab
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rituximab — One course of IV rituximab consisting of a first infusion of 1000 mg (500 mL solution) rituximab (day 1), and a second infusion of 1000 mg (500 mL solution) rituximab two weeks later (day 15)
  Arms: Rituximab
Other: Placebo — One course of IV placebo of rituximab consisting of a first infusion of 500 mL of saline (0.9% sodium chloride) infusion (day 1), and a second infusion of 500 mL of saline infusion two weeks later (day 15)
  Arms: Placebo

SUMMARY:
The main objective of the EvER-ILD2 study is to evaluate the efficacy on lung function at 6 months of one course rituximab (2 infusions) comparatively to one course of placebo (2 infusions) in a broad range of progressive ILD patients with inflammatory component.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years old
2. Who meet at least one of the following criteria for worsening ILD within 24 months:

   1. a relative decline in the FVC of >= 10% of the predicted value
   2. a relative decrease in the FVC of >=5 to 10% of the predicted value AND i) worsening respiratory symptoms OR ii) an increased extent of ILD on high-resolution CT OR iii) a relative decrease in the DLCO of >= 15% of the predicted value.
   3. worsening of respiratory symptoms AND an increased extent of ILD on high-resolution CT
3. AND presence of an inflammatory component defined by

   1. a previous histological pattern with lymphocyte infiltrations distant from pulmonary fibrosis to suggest an inflammatory component on pulmonary sample (for example: interstitial lymphoid aggregates with germinal centers, diffuse lympho-plasmocytic infiltrations, granulomas, giant cells or centrilobular inflammation…)
   2. OR a previous alveolar lymphocytosis >20% on Bronchoalveolar lavage fluid (BALF)
4. Subjects covered by the French social security system
5. Written informed consent obtained from subject
6. Ability for subject to comply with the requirements of the study

Exclusion Criteria:

1. Known diagnosis of significant respiratory disorders (asthma, tuberculosis, aspergillosis, cystic fibrosis, idiopathic pulmonary fibrosis (IPF), Connective Tissue Diseases-ILD, sarcoidosis, desquamative interstitial pneumonia, pulmonary hypertension (PAMp > 30mmHg))) or of significant severe heart failure.
2. Concomitant medical or surgical disease, clinically significant as considered by the investigator, serious or unstable, acute or chronically progressive, or any condition that could affect the safety of the patient, in the opinion of the investigator including cardiomyopathy or heart failure.
3. Patient who can not walk more than 100 meters at 6-minutes walk test
4. HRCT profile of typical usual interstitial pneumonia (UIP)
5. Histological model of typical NSIP or definitive UIP
6. Initiation of a new therapy or with interruption/modification of therapy dosage within 6 weeks prior to visit 1
7. Patient who has already received a rituximab-based treatment line
8. Known hypersensitivity to rituximab, to murine proteins or other excipients or sulfonamide antibiotics.
9. Treatment with monoclonal antibodies (such as, but not limited to, etanercept, adalimumab, efalizumab, infliximab, golimumab, certolizumab) within 6 months (if 5 half-lives ≤ 6 months) prior to inclusion.
10. Patients on a lung transplant list
11. Pregnant or breastfeeding women, or women of childbearing age not using a reliable method of contraception during the study and for 12 months following the end of the study treatment.
12. Patients at high risk of infectious complications: Human Immunodeficiency Virus (HIV) positive or other known immunodeficiency syndromes, hepatitis B and C (HBV, HCV), coronavirus disease (within 3 month) or other known viral infection, infection requiring anti-infective treatment within 4 weeks of inclusion.
13. Patients with incomplete anti-severe acute respiratory syndrome coronavirus 2 vaccine regimen (according to current recommendations) and in this case who has not receive a treatment with therapeutic antibodies anti-SARSCov2 (ex: tixagévimab/cilgavimab)
14. Patient under judicial protection, deprivation of liberty
15. Participation in other interventional research with an investigational drug or medical device.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2026-07-16 (Estimated); Study Completion 2026-07-16 (Estimated)

PRIMARY OUTCOMES:
Forced vital capacity | From baseline to 6 months
  The primary outcome is the change in Forced Vital Capacity (FVC) (in mL) from baseline to 6 months.

SECONDARY OUTCOMES:
Forced vital capacity | From baseline to 6 months
  Change from baseline to 6 months in FVC (in % of predicted)
Progression free survival (PFS) | At 6 months
  Progression free survival (PFS) defined as the time to (first event considered): a first acute exacerbation, or a relative decline in the FVC of ≥ 10% of the predicted value or the need for new immunosuppressive or/and anti-fibrotic therapies (excluding corticosteroids), or inclusion on a lung transplant list, or death.
King's Brief Interstitial Lung Disease (K-BILD) questionnaire | From baseline to 6 months
  Changes in the King's Brief Interstitial Lung Disease (K-BILD) questionnaire.15 questions about the impact of lung disease on life.
L-PF symptom questionnaire | From baseline to 6 months
  Changes in "Living Pulmonary fibrosis-symptom" questionnaire.23 questions about the impact of lung disease on life.
L-PF impact questionnaire | From baseline to 6 months
  Changes in "Living Pulmonary fibrosis-impact" questionnaire.21 questions about the impact of lung disease on life.
Cumulative doses of corticosteroids | At 6 months
  Difference in cumulative doses of corticosteroids
Diffusing capacity for carbon monoxide (DLCO) | From baseline to 6 months
  Changes in % of predicted diffusing capacity for carbon monoxide (DLCO)
6 minutes walk test | From baseline to 6 months
  Changes in the 6-minute walk test
Accelerometer-assessed physical activity | From baseline to 6 months
  Change in accelerometer-assessed physical activity
Biological analyse on markers related to B-cell depletion | From baseline to 6 months
  Changes of biological markers related to B-cell depletion
Environmental antigens | From baseline to 6 months
  Changes of serology by ELISA of 15 environmental antigens.
High-resolution computed tomography (HRCT) of chest images | From baseline to 6 months
  Changes in high-resolution computed tomography (HRCT) of chest images
Adverse events | From baseline to 6 months
  Description of All adverse events, especially serious infectious adverse events, occurring during the six-month treatment period
Pharmacokinetic parameters of rituximab | before and 2 hours after the end of each infusions, at 3 and 6 months after the first infusion
  Rituximab clearance
Pharmacokinetic parameters of rituximab | Before and 2 hours after the end of each infusions, at 3 and 6 months after the first infusion
  Volume of distribution
Pharmacokinetic parameters of rituximab | Before and 2 hours after the end of each infusions, at 3 and 6 months after the first infusion
  Half life
Severe Acute Respiratory Syndrome COronaVirus 2 (SARS COV 2) antibodies | From baseline to 6 months
  Change of SARS COV 2 antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Julien LE BONNIEC, Study Director — University Hospital Center of Tours
Locations (1):
- Chru Tours, Tours, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferreira M, Bejan-Angoulvant T, Marchand-Adam S, Mousset E, Mureau E, Jouneau S, Nunes H, Montani D, Chenivesse C, Cadranel J, Bonniaud P, Crestani B, Cottin V, Caille A; OrphaLung.. Evaluation of efficacy and safety of rituximab in patients with progressive interstitial lung disease (ILD) with inflammatory component (EvER-ILD2): A multicentre double-blind placebo-controlled randomized trial. Respir Med Res. 2025 May;87:101144. doi: 10.1016/j.resmer.2024.101144. Epub 2024 Nov 28. PMID 39693827